CLINICAL TRIAL: NCT04710524
Title: A Randomized Phase 2a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of FM101 in Adults With Nonalcoholic Fatty Liver Disease or Nonalcoholic Steatohepatitis
Brief Title: FM101 Efficacy Study in Adults With Nonalcoholic Fatty Liver Disease or Nonalcoholic Steatohepatitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Future Medicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FM101-CTP2-001
Record Dates: First submitted 2020-09-07; First posted 2021-01-14 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic Fatty Liver Disease; NAFLD; Nonalcoholic Steatohepatitis; NASH; FM101
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): orally administer placebo BID for 13 weeks except on Day 91 subject receive a single dose
  Interventions: Drug: Placebo
- FM101 150 mg BID (Experimental): orally administer FM101 150mg BID for 13 weeks except on Day 91 subject receive a single dose
  Interventions: Drug: FM101 150 mg BID
- FM101 300 mg BID (Experimental): orally administer FM101 300mg BID for 13 weeks except on Day 91 subject receive a single dose
  Interventions: Drug: FM101 300 mg BID

INTERVENTIONS:
Drug: Placebo — Placebo BID for 13 weeks
  Arms: Placebo
Drug: FM101 150 mg BID — FM101 (150 mg) BID for 13 weeks
  Arms: FM101 150 mg BID
Drug: FM101 300 mg BID — FM101 (300 mg) BID for 13 weeks
  Arms: FM101 300 mg BID

SUMMARY:
A Randomized Phase 2a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of FM101 in Adults with Nonalcoholic Fatty Liver Disease or Nonalcoholic Steatohepatitis

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the following criteria to be included in the study:

1. Be able and willing to provide written informed consent to take part in the study, and to comply with all the study's requirements.
2. Be a man or woman ≥18 years of age at screening.
3. Have c. Histologic confirmation of NASH no more than 12 months before the screening visit date, demonstrating the existence of steatosis ≥5%, hepatocyte ballooning and chronic inflammation (at least 1 point for each component), and stage 1 through stage 3 liver fibrosis according to the NASH Clinical Research Network (CRN); OR d. NAFLD based upon demonstration of at least 3 of the following 5 components of the metabolic syndrome below, at screening:

   * Fasting plasma glucose ≥100 mg/dL , or undergoing drug treatment for elevated plasma glucose concentrations
   * High-density lipoprotein-cholesterol (HDL-c) concentration <40 mg/dL in male patients, or <50 mg/dL in female patients, or undergoing drug treatment for reduced serum HDL-c concentrations
   * Serum triglyceride (TG) concentration ≥150 mg/dL, or undergoing drug treatment for elevated serum TG concentrations
   * Waist circumference >102 cm in male patients or >88 cm in female patients
   * Systolic blood pressure ≥130 mm Hg or diastolic blood pressure ≥85 mm Hg, or undergoing drug treatment for hypertension, or antihypertensive drug treatment in a patient with a history of systemic hypertension
4. Serum ALT concentration >1 × upper limit of normal (ULN) at screening
5. Undergo MRI-PDFF that demonstrates ≥8% liver steatosis during the screening period.
6. Undergo MRE with a score ≥2.9 kPa during the screening period.
7. Women of childbearing potential (WoCBP) must have a negative serum beta human chorionic gonadotropin (HCG) test result at screening.

   Female patients must agree to use highly effective birth control throughout the study and up to 30 days after the last dose of study drug has been taken. Highly effective contraception measures include the following, but not limited to:
   * Combined estrogen- and progestogen-containing hormonal contraception (oral, intravaginal and transdermal);
   * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, and implantable);
   * Intrauterine device, intrauterine hormone-releasing system, bilateral tubal, occlusion ('tubal occlusion' includes 'tubal ligation');
   * Vasectomized partner (only in the event that the vasectomized partner is the sole sexual partner of the WoCBP);
   * Sexual abstinence (defined as refraining from heterosexual intercourse) only in the event that this is the preferred lifestyle of the patient.

   Childbearing potential is defined as being fertile following menarche and until becoming postmenopausal unless permanently sterile (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).

   A postmenopausal state is defined as no menses for ≥12 consecutive months without an alternative medical cause.

   Men with partners who are WOCBP must either be surgically sterile or agree to use a barrier contraceptive for the duration of the study and up to 30 days after the last dose of study drug.
8. Be willing to maintain a stable diet, including alcohol intake this applies, and physical activity throughout the entire study.

Exclusion Criteria:

Individuals meeting any of the following criteria at screening or baseline are ineligible to participate in this study:

1. Any patient who refuses to provide written informed consent to take part in the study, and/or appears unwilling to comply with study-specific requirements.
2. Female persons who are pregnant, or are breastfeeding at screening, or who plan to become pregnant during the study.
3. Body mass index (BMI) <25 kg/m2.
4. Fibrosis-4 index (FIB-4) >2.6 at screening.
5. Any of the following laboratory test abnormalities at screening:

   1. Serum ALT and/or AST concentration >5 × upper limit of normal (ULN)
   2. Total serum bilirubin (BR) concentration >ULN; if an established diagnosis of Gilbert's syndrome exists and the direct serum BR result at screening is less than or equal to ULN the patient may participate in the study
   3. Serum albumin concentration ≤3.5 g/dL
   4. International normalized ratio (INR) ≥1.3
   5. Platelet count less than the lower limit of normal range (LLN)
   6. Creatinine clearance rate <60 mL/minute as calculated by the modification of diet in renal disease (MDRD) estimated glomerular filtration rate (eGFR) equation
   7. Positive COVID-19 polymerase chain reaction (PCR) test result at screening NOTE: Repeat testing of a given parameter or parameters that returned ineligible results, may be performed during the same screening period in consultation with the sponsor's Medical Monitor. An interval of at least 7 days should exist between receipt of the ineligible test result and re-testing.
6. Chronic liver disease other than confirmed or suspected NASH, including but not limited to the following diagnoses / entities:

   1. Chronic hepatitis B virus infection (defined by the presence of hepatitis B surface antigen at screening) and / or chronic hepatitis C virus (HCV) infection (defined by the presence of detectable HCV ribonucleic acid (RNA) antibody [anti-HCV] at screening). Patients whose anti-HCV antibody test at screening is positive, but who test negative for HCV RNA at screening will be permitted to participate in the study as long as there has been evidence of viral negativity for at least 24 months prior to screening)
   2. Autoimmune hepatitis (AIH), or confirmed overlap syndrome of AIH and either primary biliary cholangitis or primary sclerosing cholangitis.
   3. Primary biliary cholangitis, primary sclerosing cholangitis, secondary sclerosing cholangitis whatever the basis for this, e.g. chronic pancreatitis resulting in bile duct stricture formation, recurrent extrahepatic bile duct calculus formation, arterial insult resulting in bile duct stricture formation
   4. Wilson's disease, homozygous alpha-1-anti-trypsin deficiency, hemochromatosis, drug-induced liver disease
   5. Alcoholic liver disease
   6. Suspected or confirmed hepatocellular carcinoma
7. Medical, histologic, and/or imaging history of hepatic cirrhosis.
8. Clinical, endoscopic, imaging and/or laboratory manifestations of portal hypertension, such as spider nevi, splenomegaly, clinically evident ascites formation, non-bleeding gastro-oesophageal varices.
9. Known history of human immunodeficiency virus (HIV) infection.
10. Chronic use (≥12 months) of any drug known to be associated with development of NAFLD during the five years before the anticipated Day 1 visit date, e.g. amiodarone, methotrexate, systemic glucocorticoids (unless employed at physiologic replacement doses for management of confirmed adrenal insufficiency), tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement therapy, anabolic steroids (other than testosterone replacement preparations being taken at a physiologic replacement dose for management of confirmed male hypogonadism), sodium valproate, and other hepatotoxins, e.g. minocycline.
11. Use of the following medications:

    1. GLP-1 agonists, unless on a stable dose for at least 3 months prior to screening
    2. Thiazolidinediones, obeticholic acid or vitamin E at a daily dose >400 IU daily within the 6 months before screening
    3. Statin therapy and other lipid-modifying therapies must have been used at a stable dose for ≥3 months prior to screening
    4. Oral antidiabetic medication(s) (other than those specifically excluded) must have been used / taken at a stable daily dose for ≥3 months prior to screening
12. History of significant alcohol consumption, defined as an average of >20 g/day in female patients and >30 g/day in male patients, for a period of >3 consecutive months within 1 year prior to screening, hazardous alcohol use (Alcohol Use Disorders Identification Test score ≥8), or an inability to reliably quantify alcohol consumption based upon judgment of the investigator.
13. Active substance abuse within the 1 year before the screening visit date, upon the judgement of the investigator.
14. Weight change ≥7% within the 6 months prior to screening or ≥5% within the 3 months prior to screening.
15. Prior or planned (during the study period) weight reduction surgery, e.g. sleeve gastrectomy, Roux-en-Y gastrojejunostomy.
16. Type 1 diabetes mellitus by medical history.
17. Poorly controlled type 2 diabetes mellitus (this is defined as hemoglobin A1c (HbA1c) >9.5% at screening, or a patient whose oral anti-diabetic medication dosing requires adjustment >10% less than 2 months before the screening visit date.
18. Uncontrolled systemic hypertension (either treated or untreated) defined as systolic blood pressure >160 mmHg or a diastolic blood pressure >100 mmHg at screening. A retest of blood pressure, (after establishing good blood pressure control within a reasonable period of time and up to the Baseline visit) is permissible at the discretion of the Investigator.
19. Patients who demonstrate recent evidence (within 6 months of the anticipated date of the Day 1 visit) of clinically evident and significant atheromatous cardiovascular disease, e.g. unstable angina, acute coronary syndrome, myocardial infarction, cerebrovascular accident [stroke], cerebrovascular ischemia, transient ischemic attack, and / or peripheral vascular disease requiring intervention.
20. Has taken part in a clinical trial and been administered an active investigational product being evaluated for the treatment of NASH, weight reduction and / or type 2 diabetes mellitus, during the 6 months prior to the anticipated Day 1 visit date.
21. Has participated in an investigational new drug trial during the 30 days prior to screening visit date, or within 5 half-lives of an investigational agent, whichever is longer.
22. Has a confirmed diagnosis of malignancy within 5 years prior to screening, except for basal- or squamous-cell carcinoma of the skin that has been treated successfully, or cervical carcinoma in situ that has been treated successfully. Patients with a history of other malignancies that have been treated with curative intent and who have no demonstrable disease recurrence within 5 years prior to screening may also be eligible if approved following discussion with the Sponsor's Medical Monitor. Patients under evaluation for malignant disease currently are not eligible for study participation.
23. Patients who are unable to undergo MRI studies, whatever the reason for this, e.g. claustrophobia, the presence of a device or implant that would make imaging dangerous for the patient.
24. Any other condition which, in the opinion of the Investigator, would impede compliance with, hinder completion of the study, compromise the well-being of the patient, and / or interfere with the study's endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of 13 weeks of treatment with FM101 in patients with NAFLD or NASH | Day 1 through Day 106
  The number of TEAEs (frequency of occurrence, number of subjects experiencing the event)
To assess the treatment effect of FM101 on serum ALT concentrations during 13 weeks of treatment | Day 1 through Day 91
  Changes in serum ALT level

SECONDARY OUTCOMES:
To assess the effect of 13 weeks of treatment with FM101 on the change in liver stiffness (kPa) measured by magnetic resonance imaging-magnetic resonance elastography (MRI MRE) in patients with NAFLD or NASH | Day 1 through Day 91
  Change in liver stiffness on MRE

CONTACTS AND LOCATIONS:
Overall Officials: WanSeok Jeong, MBA, Study Chair — Future Medicine Co., Ltd.
Locations (12):
- Hungary (2):
  - Semmelweis Egyetem I. sz. Sebészeti és Intervenciós Gasztroenterológiai Klinika, Budapest
  - West Health Kft.,, Budapest
- Poland (5):
  - Krakowskie Centrum Medyczne sp z o.o., Krakow
  - ID Clinic Arkadiusz Pisula, Mysłowice
  - Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Medyczne K2J2, Wołomin
  - Centrum Badan Klinicznych Piotr Napora lekarze, Wroclaw
- Spain (5):
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio (HUVR), Seville
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Clnico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No